CLINICAL TRIAL: NCT05514067
Title: Electroacupuncture for Heart Protection: Clinical Application in Patients Undergoing Cardiac Bypass Surgery
Acronym: EA-CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/2028
Record Dates: First submitted 2022-05-16; First posted 2022-08-24 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Electro-Acupuncture
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will then be randomised 1:1 to receive either the EA or standard care protocols.
Masking Description: After obtaining consent, patient's study arm will be revealed via sequentially numbered, opaque, sealed and stapled envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-acupuncture (EA) arm (Experimental): Patients with stable CAD going for coronary artery bypass graft (CABG) surgery randomized to receive EA before surgery.
  Interventions: Procedure: Electro-Acupuncture
- Standard Care arm (No Intervention): Patients with stable CAD going for coronary artery bypass graft (CABG) surgery.

INTERVENTIONS:
Procedure: Electro-Acupuncture — A single application of EA at cardiac-related acupoints administered for 30 min prior to CABG surgery.
  Arms: Electro-acupuncture (EA) arm

SUMMARY:
Coronary artery disease (CAD) is the leading cause of death and disability in Singapore and worldwide. Many patients with multi-vessel CAD require surgical revascularisation by coronary artery bypass graft (CABG) surgery, and are at risk of postsurgical complications such as peri-operative myocardial injury (PMI), left ventricular dysfunction, heart failure, and death. This risk is particularly important given that the aging population, and increased prevalence of co-morbidities (diabetes, hypertension, renal failure) and complexity of cardiac surgery, mean that higher risk patients are undergoing CABG surgery. As such, new treatment strategies are required to protect the heart during CABG surgery in order to improve health outcomes in patients with CAD. In this regard, a number of animal studies have demonstrated that electroacupuncture (EA) at cardiac-related acupoints can protect the heart against the detrimental effects of acute ischaemia/reperfusion injury (IRI). However, the mechanisms underlying the beneficial effect of EA, and whether EA can protect the heart against PMI in patients undergoing CABG surgery are not known. Therefore, in this research proposal, the investigators will investigate whether EA at cardiac-related acupoints can protect the heart against PMI during CABG surgery, and the investigators will elucidate the mechanisms underlying the cardioprotective effects of EA.

DETAILED DESCRIPTION:
There are currently no effective therapies for protecting the heart against PMI during CABG surgery and therefore, new therapeutic interventions are required to reduce the magnitude of PMI, in order to preserve LV systolic function and improve health outcomes in CAD patients undergoing CABG surgery. In this regard, electroacupuncture (EA) may provide a novel treatment strategy for protecting the heart and reducing PMI during CABG surgery, and is investigated in this TCM research proposal. The magnitude of PMI can be quantified by measuring post-operative levels of serum cardiac biomarkers such CK-MB, Troponin-T, or Troponin-I, the release of which have been associated with worse clinical outcomes following CABG surgery.

This study aims to show the benefit of EA at cardiac-related acupoints in reducing injury to the heart in terms of less PMI in patients undergoing CABG surgery and also test the possibility that EA will have benefits in other organs in terms of less acute kidney injury and preserved cognitive function, given that the blood-borne humoral factors generated by EA may also be reno- and neuroprotective. As such, the findings for this research proposal will build on evidence for the safety and efficacy of EA in the clinical setting of CABG surgery for the benefit of patients with CAD. The expected clinical benefits of reducing PMI will include improvement in short term clinical outcomes in terms of preserving LV systolic function, preventing the onset of heart failure, and improving quality of life in patients undergoing CABG surgery. This study also intends to identify and assess the cardioprotective humoral factors generated by EA at cardiac-related acupoints in stable CAD and CABG patients, providing novel therapeutic strategies for cardioprotection. In this regard, the findings from this research proposal will add new knowledge in the field of EA cardioprotection.

60 stable CAD patients undergoing planned CABG surgery will be randomized to receive either EA at cardiac-related acupoints (N=30) or standard care (N=30). A single application of EA at cardiac-related acupoints will be administered for 30 min prior to surgery. For 10 recruited CABG patients administered EA, blood samples will be collected prior to and immediately following EA, and subjected to plasma proteomics analysis to identify the factor(s) which mediate EA cardioprotection. PMI will be measured as the 48-hour area under-the-curve serum high-sensitive Troponin-T. Blood samples will be taken at pre-op and 6, 12, 24, 48 hours (post-coming off cardiac bypass) for this evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable CAD undergoing planned CABG surgery on cardiopulmonary bypass using blood cardioplegia.
* Patients aged 21 years and above.

Exclusion Criteria:

* Patients with recent myocardial infarction (<30 days)
* Patients with significant hepatic dysfunction (If available, INR>2)
* Patients with significant pulmonary disease (If available, FEV1<40% predicted). - Patients with known renal failure with a GFR≤30 mL/min/1.73 m2.
* Patients recruited into another study which may impact on this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Change of Troponin-T test result from baseline to 6 hours post-op (post coming off bypass) to assess the extend of peri-operative myocardial injury (PMI) | Blood samples will be taken at pre-op and 6 hours (post coming off bypass).
  The investigators will be assessing the cardioprotective efficacy of EA at cardiac-related acupoints in terms of changing the magnitude of PMI when compared to standard care. PMI will be measured as the 48-hour area-under-the-curve serum high-sensitive Troponin-T.
Change of Troponin-T test result from 6 hours to 12 hours post-op (post coming off bypass) to assess the extend of peri-operative myocardial injury (PMI) | Blood samples will be taken at 12 hours (post coming off bypass).
  The investigators will be assessing the cardioprotective efficacy of EA at cardiac-related acupoints in terms of changing the magnitude of PMI when compared to standard care. PMI will be measured as the 48-hour area-under-the-curve serum high-sensitive Troponin-T.
Change of Troponin-T test result from 12 hours to 24 hours post-op (post coming off bypass) to assess the extend of peri-operative myocardial injury (PMI) | Blood samples will be taken at 24 hours (post coming off bypass).
  The investigators will be assessing the cardioprotective efficacy of EA at cardiac-related acupoints in terms of changing the magnitude of PMI when compared to standard care. PMI will be measured as the 48-hour area-under-the-curve serum high-sensitive Troponin-T.
Change of Troponin-T test result from 24 hours to 48 hours post-op (post coming off bypass) to assess the extend of peri-operative myocardial injury (PMI) | Blood samples will be taken at 48 hours (post coming off bypass).
  The investigators will be assessing the cardioprotective efficacy of EA at cardiac-related acupoints in terms of changing the magnitude of PMI when compared to standard care. PMI will be measured as the 48-hour area-under-the-curve serum high-sensitive Troponin-T.

SECONDARY OUTCOMES:
Any Acute Kidney Injury | Urine output will be measured over the 3 day peri-operative period to derive the AKI grade.
  The investigators will investigate the reno-protective effects of EA at cardiac-related acupoints by comparing the AKI grade following CABG surgery between the 2 study arms.
Change in Cognitive Function measure | MMSE will be conducted prior to surgery, postoperative day 3 and postoperative week 6.
  Patient cognitive function will be assessed using the Mini-Mental State Examination (MMSE) with a maximum score of 30. Higher scores reflect better outcomes.
Change in Quality of life measure | The questionnaire will be done prior to surgery, postoperative day 3 and postoperative week 6.
  The EuroQol EQ-5D Health-Related Quality of Life questionnaire will be used to assess patient quality of life. Higher score given for health state imagined reflects better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Hausenloy, PHD, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore